CLINICAL TRIAL: NCT03684174
Title: Non-Contact Air Tonometry (Topcon CT-1®) Versus Goldmann Applanation Tonometry: a Device Comparison Study
Brief Title: Non-Contact Air Tonometry (Topcon CT-1®) Versus Goldmann
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00136
Record Dates: First submitted 2018-09-17; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Glaucoma
Keywords: Tonometry
MeSH Terms: conditions — Glaucoma | interventions — Tonometry, Ocular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Intraocular pressure measurement — Pressure tip or air puff is applied on eye

SUMMARY:
In this prospective device comparison study with 58 healthy eyes, the Topcon CT-1® showed statistically significant elevated intraocular pressure measurements compared to the gold standard Goldmann application tonometry.

DETAILED DESCRIPTION:
Introduction:

Intraocular pressure (IOP) measurement is crucial in glaucoma diagnosis and treatment. We compared a non-contact air tonometer (Topcon CT-1®) with the gold standard Goldmann Applikation tonometer (GAT).

Methods:

In this prospective, mono centric device comparison study, only healthy eyes were enrolled. IOP was measured three times with the Topcon CT-1® followed by three times GAT. Mean IOP was calculated and compared with a paired t-test, a linear regression and a Bland-Altman analysis.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers who agreed to be included in the study and were able to comply with the measurement procedures

Exclusion criteria were cor-neal abnormalities (such as oedema, scars or dystrophies, astigmatism,hyperopia or myopia > 3 dioptres), a history of ocular surgery or recent(<47 weeks) ocular disorder.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Comparison of GAT with air tonometry Topcon CT1 | 7 months
  Difference in mmHg between these two devices

CONTACTS AND LOCATIONS:
Overall Officials: Pascal B Knecht, MD PD, Study Chair — University of Zurich
Locations (1):
- Augenpraxis Centerpassage, Wettingen, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon MO, Beiser JA, Brandt JD, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Kass MA. The Ocular Hypertension Treatment Study: baseline factors that predict the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):714-20; discussion 829-30. doi: 10.1001/archopht.120.6.714. PMID 12049575
- [Background] Jorge J, Gonzalez-Meijome JM, Diaz-Rey JA, Almeida JB, Ribeiro P, Parafita MA. Clinical performance of non-contact tonometry by Reichert AT550 in glaucomatous patients. Ophthalmic Physiol Opt. 2003 Nov;23(6):503-6. doi: 10.1046/j.1475-1313.2003.00139.x. PMID 14622352
- [Background] Leske MC, Heijl A, Hussein M, Bengtsson B, Hyman L, Komaroff E; Early Manifest Glaucoma Trial Group. Factors for glaucoma progression and the effect of treatment: the early manifest glaucoma trial. Arch Ophthalmol. 2003 Jan;121(1):48-56. doi: 10.1001/archopht.121.1.48. PMID 12523884
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940